CLINICAL TRIAL: NCT03851497
Title: A Multi-center Study of Deep Learning Diagnosis and Ultrasound Elastography in Opportunistic Screening of Breast Cancer
Brief Title: Application of Deep-learning and Ultrasound Elastography in Opportunistic Screening of Breast Cancer
Status: Completed | Type: Observational
Sponsor: Peking Union Medical College Hospital (Other)
Collaborators: Peking University Third Hospital (Other); Beijing Hospital (Other Government); Beijing Chao Yang Hospital (Other); Beijing Zhongguancun Hospital (Unknown); Peking University Aerospace Center Hospital (Other); Beijing Anzhen Community Health Service Center (Unknown); First Hospital of Tsinghua University (Other); Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other); The First Affiliated Hospital of Zhengzhou University (Other); Henan Provincial People's Hospital (Other); Third Affiliated Hospital of Zhengzhou University (Other); Xinxiang Central Hospital (Other); Henan Cancer Hospital (Other Government); First Hospital of China Medical University (Other); Shengjing Hospital (Other); Liaoning Cancer Hospital & Institute (Other); West China Hospital (Other); Sichuan Provincial People's Hospital (Other); Yan'an Hospital of Kunming City (Unknown); Xi'an Central Hospital (Other); Ningxia Medical University (Other); First Hospital of Shijiazhuang City (Other); Chengde Central Hospital (Other Government); Qinghai Province Cancer Hospital (Unknown); Gansu Cancer Hospital (Other); Shanghai Zhongshan Hospital (Other); Ruijin Hospital (Other); The Affiliated Hospital of Qingdao University (Other); Qingdao Central Hospital (Other); Jining First People's Hospital (Other); Linyi Tumour Hospital (Other); The First Affiliated Hospital of Shanxi Medical University (Other); The Second Affiliated Hospital of Harbin Medical University (Other); Second Hospital of Jilin University (Other); The Second Hospital of the West Coast New Area of Qingdao (Unknown); Fudan University (Other); Tongji Hospital (Other); Jiangsu Province People's Hospital (Unknown); Peking University Shougang Hospital (Other); Gansu Jiugang Hospital (Unknown)
Responsible Party: Sponsor
Other Study IDs: S-detect 2019
Record Dates: First submitted 2019-02-21; First posted 2019-02-22 (Actual); Last update posted 2021-03-26 (Actual); Status verified 2021-03

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
As the most common cancer expected to occur all over the world, breast cancer still faces with the unsatisfied diagnostic accuracy in US imaging. S-detect is a sophisticated CAD system for breast US imaging based on deep learning algorithms. E-breast is a software installed in US machines which automatically reveals tumor elastographic features. This multi-center study intends to further validate the diagnostic efficiency of S-detect and E-breast in opportunistic breast cancer screening populations in China. Our hypothesis is that S-detect and E-breast can increase the diagnostic accuracy and specificity as compared to routinely US examinations by doctors.

ELIGIBILITY:
Inclusion Criteria:

* Female over 18 years of age;
* Had breast lesions detected by ultrasound.
* No clinical symptoms such as nipple discharge, while breast lesions were not palpable.
* Received breast surgery within one week of ultrasound examination.
* Agreed to participant in this study and signed informed consent.

Exclusion Criteria:

* Patients who had received a biopsy of breast lesion before the ultrasound examination.
* Patients who were pregnant or lactating.
* Patients who were undergoing neoadjuvant treatment.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Biologically Female
Study Population: Asymptomatic female patients voluntarily asked for breast US examination in comprehensive hospitals for breast cancer screening.
Sampling Method: Probability Sample
Enrollment: 1200 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2021-01-01 (Actual); Study Completion 2021-01-01 (Actual)

PRIMARY OUTCOMES:
Benign or malignant lesions as determined by pathology | From 2019.1.1 to 2020.1.1
  The pathological diagnosis of benign or malignant lesions from surgery samples

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China